CLINICAL TRIAL: NCT03463083
Title: Evaluation of the Analgesic Effect of Dexmedetomidine Versus Fentanyl as Adjuvants to Epidural Bupivacaine in Patients Undergoing Lumbar Spine Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Mohamed, Ahmed A., M.D. (Individual); Tarek Ahmed Radwan (Unknown); Mohamed Mahmoud Mohamed (Unknown); ismaiel saied hammad (Unknown)
Responsible Party: Principal Investigator, Ahmed Abdalla, Assistant Professor of Anesthesia &I.C.U and Pain Clinic, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N-115-2017
Record Dates: First submitted 2017-12-29; First posted 2018-03-13 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Dexmedetomidine VS Fentanyl as Adjuvants to Epidural Bupivacaine in Patients Undergoing Lumbar Spine Surgeries
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine; Fentanyl

STUDY DESIGN:
Intervention Model Description: This double-blind, prospective, randomised clinically controlled study is designed to study the efficacy of epidural analgesia of dexmedetomidine and compare the analgesic effect of its epidural injection with bupivacaine versus fentanyl with bupivacaine in the post operative period of elective spine surgeries.
  To determine if the epidural route provide an acceptable analgesia in spine surgeries and avoided the need for excessive IV analgesics. Also to determine whatever dexmedetomidine or fentanyl is more better neuroaxial adjuvant regarding providing early onset and prolonged analgesia and stable cardiorespiratory parameters.
Who Masked: Participant, Care Provider
Masking Description: An online randomization program (http://www.randomizer.org) will be used to generate random list and to allocate patients into the study groups. Random allocation numbers will be concealed in opaque closed envelops. The patient and investigator assessing study outcomes will all be blinded to the study groups allocation. The study drugs will be prepared by a separate investigator not involved in outcome assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine dexmedetomidine group (Active Comparator): Group 1 (bupivacaine + dexmedetomidine (BD) group); will Receive an epidural study solution of 18 ml of 0.25% of bupivacaine hydrochloride plus 1 ml of dexmedetomidine (1 mcg/kg) plus 1 ml normal saline keeping the total volume of 20 ml in a syringe pump .
  Interventions: Drug: Dexmedetomidine; Drug: Bupivacaine
- Bupivacaine fentanyl group (Active Comparator): Group 2 (bupivacaine + fentanyl (BF) group) ; will Receive an epidural study solution of 18 ml of 0.25% bupivacaine plus 2 ml fentanyl (1 mcg/kg) keeping the total volume of 20 ml in a syringe pump .
  Interventions: Drug: Bupivacaine; Drug: Fentanyl

INTERVENTIONS:
Drug: Dexmedetomidine — All cases of spine surgery will be done under G.A with the patient in prone position. After surgery an epidural catheter will be placed through a separate skin puncture above the incision The catheter will be positioned up to 7 cm from skin entry directing downwards in the epidural space . Once the patient in the post-operative room will be noted to have pain (VAS) of>4, the study will start. A test dose of 3 ml lignocaine with adrenaline will be injected the following parameters will be noted .
  1. The pain score, by using VAS
  2. Onset of analgesia (fall of VAS<4 ).
  3. Peak level of analgesia ( VAS score 0).
  4. Duration of analgesia (once the patient asks fwith VAS>4).
  5. Monitoring of NIBP, pulse rate, respiratory rate every 30 min.
  6. Side-effects such as nausea, vomiting, respiratory depression, Motor blockade "Bromage scale>1" Also deep sedation "Ramsay sedation scale>3" , And shivering and hypotension.
  Other Names: Dexmedetomidine bupivacaine versus fentanyl bupivacaine
  Arms: Bupivacaine dexmedetomidine group
Drug: Bupivacaine — All cases of spine surgery will be done under G.A with the patient in prone position. After surgury an epidural catheter will be placed through a separate skin puncture above the incision The catheter will be positioned up to 7 cm from skin entry directing downwards in the epidural space . Once the patient in the post-operative room will be noted to have pain (VAS) of>4, the study will start. A test dose of 3 ml lignocaine with adrenaline will be injected the following parameters will be noted .
  1. The pain score, by using VAS
  2. Onset of analgesia (fall of VAS<4 ).
  3. Peak level of analgesia ( VAS score 0).
  4. Duration of analgesia (once the patient asks fwith VAS>4).
  5. Monitoring of NIBP, pulse rate, respiratory rate every 30 min.
  6. Side-effects such as nausea, vomiting, respiratory depression, Motor blockade "Bromage scale>1" Also deep sedation "Ramsay sedation scale>3" , And shivering and hypotension.
Drug: Fentanyl — All cases of spine surgery will be done under G.A with the patient in prone position. After surgury an epidural catheter will be placed through a separate skin puncture above the incision The catheter will be positioned up to 7 cm from skin entry directing downwards in the epidural space . Once the patient in the post-operative room will be noted to have pain (VAS) of>4, the study will start. A test dose of 3 ml lignocaine with adrenaline will be injected the following parameters will be noted .
  1. The pain score, by using VAS
  2. Onset of analgesia (fall of VAS<4 ).
  3. Peak level of analgesia ( VAS score 0).
  4. Duration of analgesia (once the patient asks fwith VAS>4).
  5. Monitoring of NIBP, pulse rate, respiratory rate every 30 min.
  6. Side-effects such as nausea, vomiting, respiratory depression, Motor blockade "Bromage scale>1" Also deep sedation "Ramsay sedation scale>3" , And shivering and hypotension.
  Arms: Bupivacaine fentanyl group

SUMMARY:
To determine if the epidural route provide an acceptable analgesia in spine surgeries and avoided the need for excessive IV analgesics. Also to determine whatever dexmedetomidine or fentanyl is more better neuroaxial adjuvant regarding providing early onset and prolonged analgesia and stable cardiorespiratory parameters

DETAILED DESCRIPTION:
Relieving post-operative pain of spine surgeries has become an indispensable component in anesthesiology. Various methods have been tried for the management of post-operative pain in spine surgeries out of which regional techniques are becoming most promising. The quality of regional anesthesia has been reported to improve with the addition of opioids (such as morphine, fentanyl, and sufentanil) and other drugs (such as dexmedetomidine, clonidine, magnesium sulfate, neostigmine, ketamine, and midazolam), but no drug to inhibit nociception is without associated adverse effects . α2 adrenergic agonists have both analgesic and sedative properties when used as an adjuvant in regional anesthesia. Dexmedetomidine is an S-enantiomer of medetomidine with a higher specificity for α2-adrenoreceptor (α2 : α1, 1620 : 1) compared to clonidine (α2 : α1, 220 : 1). It was first introduced into practical use as intravenous sedative after the approval of U.S. Food and Drug Administration in 1999. Since then it has been investigated as the anxiolytic, sympatholytic, and analgesic properties related to α2-adrenoceptor binding, and it is now being used as a co-analgesic drug. As adjuvant, neuroaxial administration is the appropriate route to dexmedetomidine, because the analgesic effect of α2-agonists mostly occurs at spinal level, and dexmedetomidin's high lipophilicity facilitates rapid absorption into the cerebrospinal fluid and binding to the spinal cord α2-adrenoreceptor. regional-administeration of dexmedetomidine has been shown to exert potent antinociceptive effects in animals. To date, a few studies have reported on the effects of epidural dexmedetomidine combined with local anesthetics in humans. . Administration of an α2-agonist via an intrathecal or epidural route provides an analgesic effect in postoperative pain without severe sedation. This effect is due to the sparing of supraspinal CNS sites from excessive drug exposure, resulting in robust analgesia without heavy sedation . The adverse effects of dexmedetomidine include hypotension, hypertension, nausea, bradycardia, atrial fibrillation, and hypoxia. Fentanyl is one of the short-acting narcotic analgesics with potent morphine-like action . Neuroaxial administration of lipophilic opioids such as Fentanyl and sufentanyl tends to provide a rapid onset of analgesia. Their rapid clearance from cerebrospinal fluid may limit cephalic spread and the development of certain side effects such as delayed respiratory depression

ELIGIBILITY:
Inclusion Criteria:

1. All male patients between the age group of 18 and 65 years
2. Patients of American Society of Anaesthesiologists (ASA) class I and II.
3. Patients who will undergo lumbar spine surgeries (laminectomy ± discectomy for PIVD (Prolapse of intervertebral disc), will be enrolled for this study

Exclusion Criteria:

1. All Patients below the age of 18 years and above 65 years. Also All female patient are excluded from the study.
2. Other spine surgeries rather than laminectomy, also surgeries on more than two levels.
3. Patients with haematological disease, bleeding or coagulation test abnormalities, psychiatric diseases.

4 .Patiensts with history of drug abuse, allergy to any study medication. . 4 .Patients with cervical and thoracic spine surgeries, tubercular spine , any permanent neurological disorders and vertebral deformeties such as scoliosis and spondylolisthesis.

5. Pregnant and lactating patients .

Withdrawal criteria :

Accidental Dural puncture.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Males only included in the study to abolish sex difference in pain perception which is attributed to social conditioning and to psychological factors. Also many laboratory studies of humans have described sex differences in sensitivity to noxious stimuli, suggesting that biological mechanisms underlie such difference. In addition, sex hormones influence pain sensitivity)
Enrollment: 60 (Actual)
Dates: Start 2018-03-04 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-06 (Actual)

PRIMARY OUTCOMES:
Post-operative analgesia duration assessment | 24 hours
  The duration of effective analgesia; "it is the duration of complete pain relief (zero pain) and ends by the appearance of any pain (even VAS is of one)."

SECONDARY OUTCOMES:
Post-operative assessment of pain | 24 hours
  Post-operative assessment of pain using The Visual Analogue Scale (VAS: 0= no pain and 10 = worst possible pain).
Complete sensory and motor block | 24 hours
  Time taken to achieve complete sensory and motor block
Sedation assessment | 24 hours
  Post operative assessment of sedation using modified Ramsay scale (Grade 1, Patient is anxious and agitated or restless, 2, Patient is co-operative, oriented, and tranquil, 3, Patient responds to commands only; 4, Patient exhibits brisk response to light glabellar tap or loud auditory stimulus,5, Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus,6, Patient exhibits no response )
Heart rate monitoring | 24 hours
  Perioperative hemodynamics
Mean arterial blood pressure | 24 hours
  Perioperative hemodynamics
Vomiting assessment | 24 hours
  Post-operative assessment of vomiting
Itching assessment | 24 hours
  Post-operative assessment of itching
Urine retention assessment | 24 hours
  Post-operative assessment of urine retention
Post-operative Neusea | 24 hours
  Post-operative Neusea assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abdalla Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Via scholar Gate